CLINICAL TRIAL: NCT06674863
Title: Addressing Health Literacy With a Tailored Survivorship Care Plan to Improve Access in Underserved African American Prostate Cancer Patients
Brief Title: Addressing Health Literacy With a Tailored Survivorship Care Plan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Viraj Master, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008365; NCI-2024-08650 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008365 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6368-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Localized Prostate Carcinoma; Oligometastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (standard SCP, tailored SCP) (Experimental): Patients receive standard SCP during a provider visit and a tailored SCP with a low literacy educational supplement during a structured interview over 30-60 minutes.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Questionnaire Administration; Other: Supportive Care
- Group II (standard SCP) (Active Comparator): Patients receive standard SCP using the prostate cancer ASCO template during a provider visit and undergo a structured interview over 30-60 minutes.
  Interventions: Other: Interview; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Other: Educational Intervention — Receive a low literacy educational supplement
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (standard SCP, tailored SCP)
Other: Interview — Undergo a structured interview
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive standard SCP
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
Other: Supportive Care — Receive a tailored SCP
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Group I (standard SCP, tailored SCP)

SUMMARY:
This clinical trial compares the impact of a tailored survivorship care plan (SCP) to a standard SCP on the understanding of and access to survivorship care in black or African American patients with prostate cancer that has not spread to other parts of the body (localized) or that has spread from where it first started (primary site) to a limited number of places in the body (oligometastatic). SCPs summarize treatment history and recommendations for monitoring and maintaining health, and may also include potential long term effects of treatments received. The intention of a SCP is to help patients participate in their own health care. However, many patients have below basic levels of health literacy, meaning, they have a lower ability to obtain, communicate, process and understand basic health information and services to make health decisions. In fact, poor health literacy has been linked with worse quality of life in prostate cancer survivors. A tailored SCP includes the addition of an educational supplement based on lower reading and writing skills (low literacy) and may address health literacy barriers to understanding of treatment options and side effects. A standard SCP uses a template based on the American Society of Clinical Oncology (ASCO) guidelines for prostate cancer. A tailored SCP with low literacy educational supplements may be more effective compared to a standard SCP in improving understanding and access to survivorship care in black or African American patients with localized or oligometastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare outcomes after patients receive usual care from their providers with a standard SCP and after patients receive tailoring of the SCP with the low literacy educational supplement.

II. To quantify the potential benefit of tailoring the care plan and the educational supplement.

III. Compare providers' assessment of patients':

IIIa. Health literacy; IIIb. Comprehension of survivorship care recommendations; IIIc. Understanding of long term and late effects from treatment; IIId. To measures obtained from patients.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (INTERVENTION): Patients receive standard SCP during a provider visit and a tailored SCP with a low literacy educational supplement during a structured interview over 30-60 minutes.

GROUP II (CONTROL): Patients receive standard SCP using the prostate cancer ASCO template during a provider visit and undergo a structured interview over 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Black and African American men who are disease-free after completing primary surgery and/or radiation treatment for localized or oligometastatic prostate cancer between 1 to 4 years prior to enrollment. (Race/ethnicity per medical records and self report)
* Patients who are still receiving adjuvant androgen deprivation therapy following primary radiation with non-palliative intent may be included

Exclusion Criteria:

* Dementia or cognitive impairment per provider clinical assessment
* Unable to give informed consent in the judgement of the patient's oncology provider
* Recurrent prostate cancer after primary treatment
* Less than 18 years of age at the time of informed consent
* Diagnosis of active second malignancy requiring treatment
* Individuals who are not able to clearly understand English since the outcome measures require understanding of English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehension of survivorship care recommendations and prostate specific antigen surveillance | At baseline and up to 3 month phone call
  Comprehension will be scored as dichotomous variables, correct or incorrect. The proportion of patients who correctly understand after the standard survivorship care plan (SCP) compared to the proportion who correctly understand after the standard SCP + tailoring + educational support will be analyzed using a two-tailed Z-score test for equality of two proportions at a significance level of P < 0.05.
Comprehension of treatment side effects and late effects | At baseline and up to 3 month phone call
  Comprehension will be scored as dichotomous variables, correct or incorrect. The proportion of patients who correctly understand after the standard SCP compared to the proportion who correctly understand after the standard SCP + tailoring + educational support will be analyzed using a two-tailed Z-score test for equality of two proportions at a significance level of P < 0.05.

SECONDARY OUTCOMES:
Access to survivorship care for late and long-term side effects | At baseline and up to 3 month phone call
  Will be assessed using the Patients Access Score (PAS). Descriptive statistics will be used to characterize patient access to survivorship care. The difference in mean PAS will be compared between the two arms using a 2 sample t-test. Results will be compared to previous studies, published work, and other historical cohorts. The concordance of urologists' assessment of patients' outcomes with outcomes obtained from patients will be analyzed as the percent of concordant responses, and with unweighted and weighted kappa coefficients. Linear regression models will be used to identify predictors of access to survivorship care. Parsimonious models will be favored due to the relatively small sample size.
Decision regret | At baseline and up to 3 month phone call
  Descriptive statistics will be used to characterize decision regret. Results will be compared to previous studies, published work, and other historical cohorts. The concordance of urologists' assessment of patients' outcomes with outcomes obtained from patients will be analyzed as the percent of concordant responses, and with unweighted and weighted kappa coefficients. Parsimonious models will be favored due to the relatively small sample size.
Change in decisional conflict | At baseline and up to 3 month phone call
  The two-sample t-test will be used to evaluate the change in the average decisional conflict score between patients in the control arm (standard SCP) and patients in the intervention arm (standard SCP + tailoring + educational supplement).
Preparedness for survivorship | At baseline and up to 3 month phone call
  Descriptive statistics will be used to characterize preparedness for survivorship. Results will be compared to previous studies, published work, and other historical cohorts. The concordance of urologists' assessment of patients' outcomes with outcomes obtained from patients will be analyzed as the percent of concordant responses, and with unweighted and weighted kappa coefficients. Parsimonious models will be favored due to the relatively small sample size.
Patient self-efficacy | At baseline and up to 3 month phone call
  Descriptive statistics will be used to characterize patient self-efficacy. Results will be compared to previous studies, published work, and other historical cohorts. The concordance of urologists' assessment of patients' outcomes with outcomes obtained from patients will be analyzed as the percent of concordant responses, and with unweighted and weighted kappa coefficients. Parsimonious models will be favored due to the relatively small sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Viraj Master, MD, PhD, FACS, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Atlanta, Georgia